CLINICAL TRIAL: NCT04412278
Title: Impact of COVID-19 Pandemic on Perceived Exercise Benefits and Barriers: Cross Sectional Study on Turkish Society and Interpretation With Physical Activity Level
Brief Title: Impact of COVID-19 Pandemic on Perceived Exercise Benefits and Barriers
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Begüm Okudan, MSc. Pt, Okan University
Other Study IDs: 500600127
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: COVID; Isolation, Social
Keywords: Covid 19; Physical activity level; Exercise benefits and barriers; Turkish Society; Social Isolation
MeSH Terms: conditions — Social Isolation; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Turkish society: Individuals speak Turkish and lives in Turkey, ages between 15 - 65, literate and with internet access
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — Volunteer individuals enrolled the study after approval an online informed consent form. Sociodemographic data of the participants recorded as an online survey. Then, patient reported outcomes were used to assess physical activity level (International Physical Actvity Questionairre) and Exercise Benefits and Barriers (Exercise Benefits and Barriers Scale).

SUMMARY:
It is aimed to determine the physical activity level and exercise benefits and barriers caused by Covid-19 pandemic and reveal the relationship between them.

DETAILED DESCRIPTION:
Study hypothesis that people are tend to be physically inactive while Covid-19 pandemic. It is aimed to determine the exercise benefits and barriers caused by Covid-19 pandemic and reveal the relationship among gender, age, marial status and physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* being Turkish
* understanding Turkish
* being between the age of 15 - 65
* being literate
* have internet access

Exclusion Criteria:

* having a disable condition to exercise
* having missing value on outcome measures
* giving incomprehensible answering

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of the individuals between 15 - 65 ages in Turkey is 56.391.925 people. It is calculated that there are 42.463.119 individuals cover the criterion as universe of the study.
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Exercise Benefits and Barriers Scale | three months after Covid 19 recognised as pandemic
  The Exercise Benefits/Barriers Scale (EBBS) was developed in response to a need for an instrument to determine perceptions of individuals concerning the benefits of and barriers to participating in exercise. The instrument may be scored and used in its entirety or as two separate scales. The instrument has a four-response, forced-choice Likert-type format with responses ranging from 4 (strongly agree) to 1 (strongly disagree). Scores on the total instrument can range from 43 to 172. The higher the score, the more positively the individual perceives exercise. When the Benefits Scale is used alone, the score range is between 29 and 116. When the Barriers Scale is used alone, scores range between 14 and 56. If used alone, the Barriers Scale does not need to be reverse-scored. In this instance, the higher the score on the Barriers Scale, the greater the perception of barriers to exercise.
Sociodemographic information | three months after Covid 19 recognised as pandemic
  Participants will be asked to give information about: age, gender, educational status, height, weight, occupation, working status, whether they have a chronic disease.

SECONDARY OUTCOMES:
International Physical Activity Questionairre | three months after Covid 19 recognised as pandemic
  The IPAQ-S developed for participants to report activities performed for at least 10 minutes during the last 7 days. Respondents will be asked to report time spent in physical activity performed across leisure time, work, domestic activities, and transport at each of 3 intensities: walking, moderate, and vigorous. Using the instrument's scoring protocol total weekly physical activity was estimated by weighting time spent in each activity intensity with its estimated metabolic equivalent (MET) energy expenditure. The IPAQ scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively. Participants will be considered to have met American Collage of Sports Medicine physical activity recommendations. if they reported at least 150 min/wk of walking, moderate, or vigorous intensity physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data wil be stored by researches, if needed for scientific purposes, it can be discussed to share .